CLINICAL TRIAL: NCT00468208
Title: A Multi-Center, Open-label Pilot Study of Abatacept (CTLA4-Ig) in the Treatment of Mild Relapsing Wegener's Granulomatosis
Brief Title: Abatacept in Treating Adults With Mild Relapsing Wegener's Granulomatosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDCRN 5522; U54AR057319 (NIH)
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-12

CONDITIONS: Wegener's Granulomatosis
Keywords: Vasculitis; Relapse; Wegener's; Treatment
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Vasculitis; Recurrence | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants will receive abatacept intravenously at study visits on Days 1, 15, and 29, and then once a month thereafter.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — A participant's abatacept dose depended on body weight and will remain the same throughout the study:
  * 500 mg of abatacept for body weight less than 60 kg
  * 750 mg of abatacept for body weight between 60 and 100 kg
  * 1000 mg of abatacept for body weight greater than 100 kg
  Abatacept is administered in a 30-minute intravenous infusion.

SUMMARY:
Wegener's granulomatosis (WG) is a rare disease that causes inflammation of blood vessels, or vasculitis. It may involve many different parts of the body, but typically affects the upper and lower respiratory tract and kidneys. The purpose of this study is to determine the safety and effectiveness of the medication abatacept in treating adults with mild relapsing WG.

DETAILED DESCRIPTION:
Current standard treatment for WG involves various medications and is based on disease severity. Unfortunately, more than 50% of people experience a relapse after remission, placing them at risk for additional organ damage and medication toxicity. To prevent this, safer and more effective treatments for mild relapses are needed. Several studies have shown that activated T cells, a type of white blood cell important in regulating immune responses, play a role in WG. Abatacept, an immunoglobulin-based medication approved by the FDA to treat rheumatoid arthritis, acts by preventing T-cell activation and may be useful in treating mild relapses of WG. The purpose of this study is to determine the safety and effectiveness of abatacept in treating adults with mild relapsing WG.

Participants will receive abatacept intravenously at study visits on Days 1, 15, and 29, and then once a month thereafter. A participant's abatacept dose is based on body weight and will remain the same throughout the study. Participants who are receiving maintenance immunosuppressive medications consisting of methotrexate, azathioprine, or mycophenolate mofetil at the time of enrollment will remain on these medications without dosage increase or reduction. Eligible participants may be on up to prednisone 15mg daily at the time of relapse. Following the development of relapse, participants may be treated with up to prednisone 30mg daily if necessary, but must to be back to the same dose that they had been on prior to relapse by Month 2. All study visits include medication review, physical exam, blood and urine collection, and questionnaires. A chest x-ray, computed tomography (CT) scan of the chest and sinuses, and lung function testing will occur at some study visits. Participants whose symptoms did not improved by Month 2 will be taken off abatacept. Any participants undergoing early termination or, after common closing, will undergo three follow-up study visits at 1, 3, and 6 months after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of WG, meeting at least 2 of the 5 modified American College of Rheumatology (ACR) criteria. More information about this criterion can be found in the protocol.
* Relapse of WG within the past 28 days where disease activity is confined to one or more of the following sites and where the symptoms/signs are of such a nature that the usual treatment would consist of the reinstitution or increase in GC to no more than prednisone 30mg daily and/or an increase or addition of a second immunosuppressive agent other than CYC (more specific information about this criterion can be found in the protocol):

  1. Sinonasal disease
  2. Oral mucosa ulceration
  3. Skin disease
  4. Musculoskeletal disease
  5. Pulmonary parenchymal disease
  6. Mild ocular disease
  7. Subglottic inflammation without significant stenosis
  8. Otic disease
  9. Breast involvement
  10. Urogenital involvement
  11. Other mild disease
* Age of 15 years or older
* Willing and able to undergo treatment and attend follow-up visits
* Willing to use effective forms of contraception throughout the study

Exclusion Criteria:

* Disease involvement that does not meet the criteria for mild disease. More information about this criterion can be found in the protocol.
* Disease activity that would usually be treated first with cyclophosphamide
* Presence of disease activity for which the investigator would normally treat the participant with more than prednisone 30 mg daily.
* Receiving cyclophosphamide at study entry
* Treatment with prednisone at a dose of more than 15 mg daily at the time of relapse. Subjects will be eligible if prednisone was initiated or dose increased in the period between relapse and study enrollment provided that the prednisone dose was 15 mg daily or less at the time when the relapse occurred, the prednisone dosage was increased no higher than 30 mg daily following the recognition of relapse, and that the dosage increase was made no more than 28 days prior to enrollment.
* Active infection
* HIV infected, hepatitis C virus infected, or positive for hepatitis B
* Unable to follow through with study participation
* Cytopenia, defined as platelet count less than 80,000/mm3, absolute neutrophil count less than 1500/mm3, OR hematocrit less than 20%
* Kidney insufficiency
* Use of illegal drugs
* Any other uncontrolled disease that would prevent participation
* History of cancer. More information about this criterion can be found in the protocol.
* Received an investigational medication or procedure within 30 days of study entry
* Received a live vaccine within 4 weeks of study entry
* Positive tuberculin skin test. More information about this criterion can be found in the protocol.
* Tuberculosis as indicated by radiographic evidence
* Past treatment with rituximab within the past 12 months, or past treatment with rituximab more than 12 months ago where the B lymphocyte count has not returned to normal
* Certain other diseases. More information about this criterion can be found in the protocol.
* Pregnant or breastfeeding

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol A. Langford, MD, MHS, Principal Investigator — The Cleveland Clinic; Peter A. Merkel, MD, MPH, Principal Investigator — Boston University
Locations (4):
- United States (4):
  - The Johns Hopkins Vasculitis Center, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Background] Genovese MC, Becker JC, Schiff M, Luggen M, Sherrer Y, Kremer J, Birbara C, Box J, Natarajan K, Nuamah I, Li T, Aranda R, Hagerty DT, Dougados M. Abatacept for rheumatoid arthritis refractory to tumor necrosis factor alpha inhibition. N Engl J Med. 2005 Sep 15;353(11):1114-23. doi: 10.1056/NEJMoa050524. PMID 16162882
- [Background] Langford CA, Talar-Williams C, Barron KS, Sneller MC. Use of a cyclophosphamide-induction methotrexate-maintenance regimen for the treatment of Wegener's granulomatosis: extended follow-up and rate of relapse. Am J Med. 2003 Apr 15;114(6):463-9. doi: 10.1016/s0002-9343(03)00077-9. PMID 12727579
- [Background] Wegener's Granulomatosis Etanercept Trial (WGET) Research Group. Etanercept plus standard therapy for Wegener's granulomatosis. N Engl J Med. 2005 Jan 27;352(4):351-61. doi: 10.1056/NEJMoa041884. PMID 15673801
- [Result] Langford CA, Monach PA, Specks U, Seo P, Cuthbertson D, McAlear CA, Ytterberg SR, Hoffman GS, Krischer JP, Merkel PA; Vasculitis Clinical Research Consortium. An open-label trial of abatacept (CTLA4-IG) in non-severe relapsing granulomatosis with polyangiitis (Wegener's). Ann Rheum Dis. 2014 Jul;73(7):1376-9. doi: 10.1136/annrheumdis-2013-204164. Epub 2013 Dec 9. PMID 24323392
- See also: Cleveland Clinic Center for Vasculitis Care and Research website — http://my.clevelandclinic.org/rheumatology_immunology/vasculitis_center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in February 2008 and the final subject was enrolled in June 2010. Subjects were recruited through the clinical practices of each site investigator.
Pre-assignment Details: At a screening visit, participants underwent procedures to establish inclusion/exclusion criteria and then signed the informed consent form.
Groups:
- Open-label Abatacept: Participants received abatacept intravenously at study visits on Days 1, 15, and 29, and then once a month thereafter until common closing or early termination.
  Abatacept : A participant's abatacept dose was based on body weight and remained the same throughout the study:
  * 500 mg of abatacept for body weight less than 60 kg
  * 750 mg of abatacept for body weight between 60 and 100 kg
  * 1000 mg of abatacept for body weight greater than 100 kg
  Abatacept was administered in a 30-minute intravenous infusion.
Period: Overall Study
Arm/Group | Open-label Abatacept
Started | 20
Completed | 20 (All patients reached common closing or early termination)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Abatacept
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 17
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Safety of Abatacept - Number of Participants With Adverse Events
Description: This study examined the safety profile of this agent when used in Wegener's granulomatosis. Information was gathered on all adverse events with specific events being identified in the protocol for analysis that included the following:
  * Infection
  * Infusion reactions
  * Cytopenias
  * Transaminase elevation
  * Skin reactions
  * GI side effects
  * Malignancy
  All adverse events were reportable for this study.
Time Frame: Measured continuously from the screening visit through to the 6 month post-treatment study visit, up to 3 years and 4 months.
Population: This study intended to examine safety and to explore preliminary signal for efficacy of abatacept in Wegener's granulomatosis. The sample size of 20 was based upon a sufficient number of subjects to begin such pilot explorations.
Measure: Number; unit: participants
Arm/Group | Open-label Abatacept
Number analyzed (Participants) | 20
participants
  Serious adverse events | 7
  Non-serious adverse events | 16
  Infection | 14
  Infusion related (systemic) | 1
  Infusion related( intravenous site reaction) | 1
  Cytopenia | 4

2. Secondary Outcome: Disease Remission
Description: Disease remission was measured by a Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG) of 0.
  The BVAS/WG is a validated disease activity index. The BVAS/WG is designed to document new or worsening clinically active vasculitis and consists of a set of items divided into nine organ based systems. BVAS/WG scores range from 0 to 63.
Time Frame: Measured monthly until common closing or early termination,up to 3 years and 4 months.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Open-label Abatacept
Number analyzed (Participants) | 20
participants | 16

3. Secondary Outcome: Disease Improvement
Description: Disease improvement was measured by a reduction in the Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG).
  The BVAS/WG is a validated disease activity index. The BVAS/WG is designed to document new or worsening clinically active vasculitis and consists of a set of items divided into nine organ based systems. BVAS/WG scores range from 0 to 63.
Time Frame: Measured monthly until common closing or early termination, up to 3 years and 4 months.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Open-label Abatacept
Number analyzed (Participants) | 20
participants | 18

4. Secondary Outcome: Meeting Common Closing
Description: The number of subjects that reached the common closing date.
Time Frame: Number assessed at the time of common closing, up to 3 years and 4 months.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Open-label Abatacept
Number analyzed (Participants) | 20
participants | 14

5. Secondary Outcome: Disease Relapse
Description: Disease relapse was measured by a rise in the Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG) of greater than or equal to 1 after achieving remission.
  The BVAS/WG is a validated disease activity index. The BVAS/WG is designed to document new or worsening clinically active vasculitis and consists of a set of items divided into nine organ based systems. BVAS/WG scores range from 0 to 63.
Time Frame: Measured monthly until common closing or early termination, up to 3 years and 4 months.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Open-label Abatacept
Number analyzed (Participants) | 20
participants | 3

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for subjects from time of signed consent through common close out of the study. The total timeframe of adverse event collection for the study was 3 years, 3 months.
Description: All serious adverse events related to study participation were reported and were recorded and graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) manual v3.0.
Arm/Group | Open-label Abatacept
Serious Adverse Events (participants affected / at risk) | 7/20
Other Adverse Events (participants affected / at risk) | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Abatacept (N=20)
Infection - Dental (Infections and infestations) | 1 (1)
Infection - Ocular (Infections and infestations) | 2 (2)
Infection - Lung (Infections and infestations) | 1 (2)
Infection - Upper airway (Infections and infestations) | 1 (1)
Infection - Gastrointestinal (Infections and infestations) | 1 (1)
Obstruction/stenosis of airway (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Hospitalization for dilation of subglottic stenosis related to damage from granulomatosis with polyangiitis (Wegener's)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Abatacept (N=20)
Allergy/immunology - Allergic reaction/hypersensitivity (Immune system disorders) | 1 (9)
Allergy/immunology (Immune system disorders) | 1 (1)
Auditory/Ear (Ear and labyrinth disorders) | 1 (1)
Auditory/Ear - Otitis (Ear and labyrinth disorders) | 1 (1)
Blood/Bone marrow - Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Blood/Bone marrow - Leukocytes (Blood and lymphatic system disorders) | 2 (2)
Blood/Bone marrow - Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 5 (10)
Dermatology/Skin - Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatology/Skin - Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Endocrine - Thyroid function high (Endocrine disorders) | 1 (1)
Endocrine - Thyroid function low (Endocrine disorders) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 2 (2)
Gastrointestinal - Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Mucositis/stomatitis (Gastrointestinal disorders) | 1 (1)
Infection - Other (Infections and infestations) | 4 (5)
Infection - Abdomen (Infections and infestations) | 1 (1)
Infection - Bronchus (Infections and infestations) | 2 (2)
Infection - Lung (Infections and infestations) | 1 (1)
Infection - Middle ear (Infections and infestations) | 1 (1)
Infection - Nose (Infections and infestations) | 1 (1)
Infection - Sinus (Infections and infestations) | 1 (1)
Infection - Skin (Infections and infestations) | 1 (1)
Infection - Soft tissue (Infections and infestations) | 1 (1)
Infection - Stomach (Infections and infestations) | 2 (2)
Infection - Upper airway (Infections and infestations) | 3 (5)
Infection - Urinary tract (Infections and infestations) | 1 (1)
Metabolic/Laboratory - Creatinine (Metabolism and nutrition disorders) | 1 (1)
Metabolic/Laboratory - Glucose high (Metabolism and nutrition disorders) | 1 (6)
Metabolic/Laboratory - Sodium high (Metabolism and nutrition disorders) | 1 (1)
Metabolic/Laboratory - Triglyceride high (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 4 (4)
Ocular/Visual - Other (Eye disorders) | 1 (1)
Ocular/Visual - Vision blurred (Eye disorders) | 1 (1)
Ocular/Visual - Vision photophobia (Eye disorders) | 1 (1)
Ocular/Visual - Watery eye (epiphora, tearing) (Eye disorders) | 2 (2)
Pain - Back pain (General disorders) | 1 (1)
Pulmonary/Upper respiratory (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pulmonary/Upper respiratory - Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The main limitation of this trial is the small sample size and the open-label, uncontrolled design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No